CLINICAL TRIAL: NCT05310617
Title: Parental Project and Premature Ovarian Insufficiency
Acronym: ParentIOP
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220208
Record Dates: First submitted 2022-03-21; First posted 2022-04-05 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Primary Ovarian Insufficiency; Infertility
Keywords: spontaneous pregnancy; adoption; oocyte donation; parental project
MeSH Terms: conditions — Primary Ovarian Insufficiency; Infertility | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — Survey on the parental project and its realisation

SUMMARY:
One of the main repercussions of POI is infertility. When the diagnosis of POI is announced, the question of fertility is addressed and the patient is often directed towards egg donation or adoption when she has a parental project. However, there are cases of spontaneous pregnancies after diagnosis.

This study was conducted to determine the proportion of patients with POI who were able to realize a parental project after diagnosis in the long term and by what means.

DETAILED DESCRIPTION:
The investigators propose to study patients with POI who were hospitalized in the endocrinology and reproductive medicine department of the Pitié-Salpêtrière Hospital for the etiological assessment of ovarian failure and its consequences between December 31, 1982 and January 12, 2021. The investigators will only include patients who were admitted to the day hospital because we have a complete etiological workup and a complete history for them, which allows investigators to describe the population properly. The patients must be over 18 years old at the time of the survey in order to be able to evaluate the presence of a parental project only in adult patients.

Patients for whom there is no valid contact information in the computer file (postal address or valid email address or cell phone number) or whose last consultation was more than 2 years ago will be excluded. Patients with Turner syndrome will be excluded because they may have comorbidities, particularly cardiac, that contraindicate pregnancy. Patients with POI secondary to oncological treatments (gonadotoxic chemotherapy or pelvic radiotherapy) will also be excluded because of the uncertain prognosis and the contraindications to pregnancy in case of hormone-dependent tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years old at the time of the survey
* Patients with a diagnosis of PIO according to the current definition: cycle disturbances of more than 4 months and FSH > 25 on 2 measurements one month apart
* Patients having been hospitalized in day hospital (HDJ) in the endocrinology and reproductive medicine department of the Pitié-Salpêtrière hospital for the etiological assessment of ovarian insufficiency and its repercussions between December 31, 1982 and January 12, 2021
* Valid contact information available: address, cell phone, e-mail
* Patients who have been informed and do not object to participate in the study

Exclusion Criteria:

* Turner syndrome
* POI secondary to oncology treatments (chemotherapy, pelvic radiotherapy)
* Opposition to participating in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients with POI who were hospitalized in a day hospital (HDJ) in the endocrinology and reproductive medicine department of the Pitié-Salpêtrière hospital for the etiological assessment of ovarian insufficiency and its repercussions between 31/12/1982 and 12/01/2021
Sampling Method: Non-Probability Sample
Enrollment: 324 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
Realisation of parental project | data from patients with a diagnosis between 31/12/1982 and 12/01/2021 and whose opposition to the study is not expressed
  Determine proportion of patient who realised a parental project after the diagnosis of POI

SECONDARY OUTCOMES:
Determine how and to what extent they have carried out their parental project | data from patients with a diagnosis between 31/12/1982 and 12/01/2021 and whose opposition to the study is not expressed
  Evaluation if, after the diagnosis of POI, the parental project was realized through: spontaneous pregnancy or egg donation, simple stimulation or in vitro fertilization, embryo reception, or the adoption of a child after the diagnosis of POI
determine how many children on average these patients had after the diagnosis of POI. | data from patients with a diagnosis between 31/12/1982 and 12/01/2021 and whose opposition to the study is not expressed
  Evaluation of the number of children born after the diagnosis of POI
determine the delay between the diagnosis of POI and the birth of the first child after the diagnosis according to the method | data from patients with a diagnosis between 31/12/1982 and 12/01/2021 and whose opposition to the study is not expressed
  Evaluation of the time between the diagnosis of POI and the birth of the first child after diagnosis according to the method (egg donation, spontaneous pregnancy, adoption, etc.)
Survey. Describe the characteristics of patients who were able to have a child after diagnosis | data from patients with a diagnosis between 31/12/1982 and 12/01/2021 and whose opposition to the study is not expressed
  Evaluation of the characteristics of patients who were able to have a child after diagnosis:
  o age at diagnosis
Survey. Describe the characteristics of patients who were able to have a child after diagnosis | data from patients with a diagnosis between 31/12/1982 and 12/01/2021 and whose opposition to the study is not expressed
  Evaluation of the characteristics of patients who were able to have a child after diagnosis:
  o AMH level
Survey. Describe the characteristics of patients who were able to have a child after diagnosis | data from patients with a diagnosis between 31/12/1982 and 12/01/2021 and whose opposition to the study is not expressed
  Evaluation of the characteristics of patients who were able to have a child after diagnosis:
  o FSH level
Survey. Describe the characteristics of patients who were able to have a child after diagnosis | data from patients with a diagnosis between 31/12/1982 and 12/01/2021 and whose opposition to the study is not expressed
  Evaluation of the characteristics of patients who were able to have a child after diagnosis:
  o presence of follicles on ultrasound
Survey. Describe the characteristics of patients who were able to have a child after diagnosis | data from patients with a diagnosis between 31/12/1982 and 12/01/2021 and whose opposition to the study is not expressed
  Evaluation of the characteristics of patients who were able to have a child after diagnosis:
  o cause of POI
Survey. Describe the characteristics of patients who were able to have a child after diagnosis | data from patients with a diagnosis between 31/12/1982 and 12/01/2021 and whose opposition to the study is not expressed
  Evaluation of the characteristics of patients who were able to have a child after diagnosis:
  o number of pregnancies prior to diagnosis
Survey. Describe the characteristics of patients who were able to have a child after diagnosis | data from patients with a diagnosis between 31/12/1982 and 12/01/2021 and whose opposition to the study is not expressed
  Evaluation of the characteristics of patients who were able to have a child after diagnosis:
  o number of children before diagnosis
Survey. Describe the characteristics of patients who were able to have a child after diagnosis | data from patients with a diagnosis between 31/12/1982 and 12/01/2021 and whose opposition to the study is not expressed
  Evaluation of the characteristics of patients who were able to have a child after diagnosis:
  o normal puberty
Survey. Describe the characteristics of patients who were able to have a child after diagnosis | data from patients with a diagnosis between 31/12/1982 and 12/01/2021 and whose opposition to the study is not expressed
  Evaluation of the characteristics of patients who were able to have a child after diagnosis:
  o age at menarche

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Touraine, Pr, Principal Investigator — APHP
Locations (1):
- Service d'endocrinologie et médecine de la reproduction, Paris, France

IPD SHARING:
Plan to Share IPD: No